CLINICAL TRIAL: NCT03012152
Title: A Comparative Study Between Oncoplastic Breast Surgery and Standard Conservative Surgery:Margin Status and Patient Satisfaction Among Egyptian Females
Brief Title: A Comparative Study Between Oncoplastic Breast Surgery and Standard Conservative Surgery:Margin Status and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abdel-samii, Lecturer of General surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16379
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Breastcancer
Keywords: Oncoplastic surgery; Standard conservative surgery; Patient satisfaction; Margin Status
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard conservative group (Active Comparator): Group A (35 patients) have standard curative conservative breast surgery without integration of plastic techniques .
  .
  Interventions: Procedure: Standard conservative breast surgery
- Oncoplastic group (Active Comparator): Group B(35 patients) have curative oncoplastic surgery in which plastic techniques integrated with oncological procedures
  Interventions: Procedure: Oncoplastic breast surgery

INTERVENTIONS:
Procedure: Standard conservative breast surgery
  Arms: Standard conservative group
Procedure: Oncoplastic breast surgery
  Arms: Oncoplastic group

SUMMARY:
This non randomized study is a comparative study between standard conservative breast surgery and oncoplastic surgery as regard margin status and patient satisfaction.

DETAILED DESCRIPTION:
This planned study was conducted on 70 female patients presented to our tertiary referral breast unit at Ain Shams University hospitals with breast cancer amid the period from September 2012 to May 2013 .

Every one of them signed an informed consent to partake in this study that was approved in a meeting held by the ethical committee on august 2012 at Ain Shams University. All patients sharing in the study received closed envelope before surgery in a randomized way in which the surgical technique is written either standard conservative surgery or oncoplastic surgery(Double Blind).

Our patients were partitioned into 2 equal groups: group A (35patients) who underwent standard conservative surgery, group B (35patients) who underwent oncoplastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients with stage 1,2 breast cancer.

Exclusion Criteria:

* Patients >60 years.
* Patients with previous breast surgery.
* patients candidate for mastectomy or palliative excision. Patients with collagen disease.

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Margins in all specimens measured in millimeters 2. | 2 years

IPD SHARING:
Plan to Share IPD: Undecided